CLINICAL TRIAL: NCT02578927
Title: Green Tea Attenuates Pressure Reduction Induced by a Session of Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Manoel Miranda Neto, Graduate, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FUParaíba
Record Dates: First submitted 2015-09-11; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GT+Ex (Experimental): Ingestion of one dose of 2 g of green tea (GT) ingested at 10 minutes after the period of rest. After the Ingestion, the volunteers practice aerobic exercise (EX) in treadmill.
  Interventions: Dietary Supplement: GT+Ex
- PL+Ex (Placebo Comparator): Ingestion of one dose 2 g of placebo (PL) ingested at 10 minutes after the period of rest. After the Ingestion, the volunteers practice aerobic exercise (EX) in treadmill.
  Interventions: Dietary Supplement: PL+Ex
- Green Tea (Active Comparator): Ingestion of one dose 2g of green tea (GT) at 10 minutes after the period of rest. In this section the volunteers does not practice aerobic exercise.
  Interventions: Dietary Supplement: Green Tea

INTERVENTIONS:
Dietary Supplement: GT+Ex — In this session the volunteers ingested capsules with 2g of powder green tea before exercise
  Arms: GT+Ex
Dietary Supplement: PL+Ex — In this session the volunteers ingested capsules with 2g of placebo before exercise
  Arms: PL+Ex
Dietary Supplement: Green Tea — In this investigation the volunteers ingested capsules with 2g of powder green tea before the rest similar to the exercise time
  Arms: Green Tea

SUMMARY:
The objective is to investigate whether the ingestion of green tea prior to physical exercise improvement post-exercise hypotension (PEH). Double-blind, randomized, placebo study. Fifteen hypertensive (53±4.5 years) performed three procedures: green tea+exercise (GT+Ex), placebo+exercise (PL+Ex), green tea without exercise (GT). Thirty minutes after ingesting 2g of green tea or placebo, they performed treadmill walking (60 minutes), 60 to 85% of maximum heart rate intensity in procedures with exercises. BP was measured at rest and at every 10 minutes after exercise (60 minutes). Blood samples were taken before the ingestion of green tea or placebo and immediately after exercise to determine Malondialdehyde (MDA) and Nitrite (NO) dosages. Reduction of systolic BP compared with the rest, during PL+Ex recovery procedure.

DETAILED DESCRIPTION:
Subjects of study: Double- blind study, randomized and placebo, conduced with fifteen both sexes hypertensive individuals, physically active and practitioners of exercises for at least 3 months prior to trials. All patients were users of anti- hypertensive medication except beta- blockers and maintained medication throughout study period. They were demanded not to be diabetic and women not menopaused. The research was approved by the Ethics Committee on Research with Human Beings of the Health Sciences Centre at the Federal University of Paraiba- CEP/ CCS, under the protocol 0120/13. Individuals were required to sign The Free and Clarified Consent Term (FCCT), according to resolution 196/96 of National Health Council.

Study Designs: subjects performed three experimental procedures, two practicing aerobic exercises and one without physical exercises. The sessions with exercises were conducted under previous administration of a green tea dosage or placebo (GT+Ex or PL+Ex), ingested 30 minutes before the start of exercises protocol. In the session without exercises (GT) they ingested green tea and remained sit during the same period destined to the exercises. Heart Rate Measurement were registered at rest (RHR) and in every ten minutes during physical exercise protocol. BP measurements were taken before (at rest), immediately after exercise and in every ten minutes during a recovery period of 60 minutes after the end of exercise protocol, or in the period they remained sit. Blood samples were collected prior and immediately after exercise or period without exercise for analysis of plasmatic concentration of anti and pro- oxidant agents (nitrite- NO and Malondialdehyde- MDA).

Instruments and Procedures:Physical Exercises: After the purposes of the research were clarified to the individuals, they were invited to proceed to the laboratory in order for exercise sessions performance. The groups were submitted to three sessions, two of those on treadmill aerobic exercise during 60 minutes. Furthermore, it was established that the individuals should practice exercises scoring between 11 and 14 in Borg and Noble's Subjective Perceived Exertion Scale. They were requested to hold the intensity of physical exercises from 60% to 85% of HRmax (maximum Heart Rate), monitored during sessions with a Polar frequency meter model RS800CX (Polar ElectroOy, Kempele, Finland).

Supplementation of Green Tea or Placebo: Green tea and placebo capsules were produced in a compounding laboratory. The investigators used 2g of green tea dried leaves and discovered an improvement in oxidative stress. The group with green tea consumption ingested capsules with 2g of concentrated powder, approximately 1960mg in polyphenols (636mg of epigallocatechin gallate) and 20mg of caffeine; placebo group consumed capsules containing 2g of cornstarch powder, all swallowed with water. Capsules were administered to patients after a skilled professional collected blood samples. Researchers conducted supplementation of substances after pre- exercise blood collection and sessions initiated only 30 minutes after the ingestion of capsules, which is the time required by the body to absorb nutrients.

Blood Pressure Measurement: Individuals had their BPs checked previously, immediately after the end of the exercise and during 60 minutes post- exercise. BP at rest was verified after the subjects remained sit for 10 minutes. By the end of the walking session, BP was checked with sitting subjects. During recovery, BP was verified in every 10 minutes during all 60 minutes of walking session. The protocol adopted was the one proposed by the Brazilian Society of Cardiology and the Brazilian Society of Hypertension.

Blood Collection Protocol: Performed prior and immediately after exercise. Ten milliliters (ml) of blood were collected from the antecubital vein, of which five ml were placed in test tubes containing EDTA and carefully homogenized by inversion. The other five ml were placed in tubes without any anticoagulant. Then they were centrifuged at 1500 rpm for 20 minutes. Plasma was isolated, placed in ependorf tubes and refrigerated in 20 ºC until analysis.

Evaluation of oxidative stress (MDA): Oxidizing activity was quantified through thiobarbituric acid reaction with the products from hydroperoxides decomposition. Therefore, 250 µl of sample was added to KCl and incubated in water bath maintained at 37° C for 60 minutes. Then mixture was precipitated with 35% AA perchloric and centrifuged at 14000 rpm and 4°C for 10 minutes. Supernatant was transferred to new ependorfs, adding 400 µl of 0.6% thiobarbituric acid and incubated at 95-100° C for 30 min. After cooling, material was read by spectrophotometer at a wavelength of 532nm.

Nitrite Dosage The method was based on the Griess reagent usage. Reagent was prepared utilizing equal parts of 5% phosphoric acid, 0.1% N-1-naphthalenediamine (NEED), 1% sulphanilamide, 5% in phosphoric acid and distilled water. To accomplish the test, 100 µl of 10% homogenate supernatant made with potassium phosphate buffer was added to 100µl Griess reagent. Regarding the white one, 100 µl reagent was added to 100 µl of buffer and series of dilutions were conducted to obtain standard curve (100, 50, 25 12.5, 6.25, 3.12, 1.56 µm) of nitrite. The entire test was executed in a 96 well- plate template with reader at an absorbance range of 560 nm.

Data Analysis Process: Initially, all data were tested concerned its normality and variability in standard error. Subsequently, one-way ANOVA tests were applied in order to compare basal conditions within three days of proceedings. Instat 3.0 software (GraphPAdInstat, San Diego, CA, USA) was utilized during analysis.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive
* Physically active for at least 3 months
* Not diabetics individuals.

Exclusion Criteria:

* Modifying the therapeutic treatment during the study
* Use beta-blocker drugs, and calcium channel blockers
* Menopausal women.

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Change from baseline Bood Pressure at 60 minutes post exercise in the same experimental session
  The sessions of exercise were released with interval of 30 days between them, thus each volunteer devoted an average 40 days to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Manoel Miranda Neto, graduation, Principal Investigator — Federal University of Paraíba